CLINICAL TRIAL: NCT00752076
Title: Detection of Epithelial Growth Factor Receptor (EGFR) Mutation in Malignant Pleural Effusion of Lung Cancer Patients and Cancer Cell Lines Establishment
Brief Title: Detection of EGFR Mutation in Malignant Pleural Effusion of Lung Cancer Patients and Cancer Cell Lines Establishment
Acronym: EGFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Department of Internal Medicine, National Taiwan University Hospital, Chest medicine devision
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200804019R
Record Dates: First submitted 2008-09-10; First posted 2008-09-15 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: NSCLC
Keywords: EGFR mutation; NSCLC cell line; Malignant pleural effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): We collected malignant pleural effusion for NSCLC cell lines with different EGFR mutations development and then we can compare the difference responses and signal pathways in these cell lines. We can also explore the detailed mechanism of TKI responsive cancer cell and try to develop other agent to enhance the pathways.
  Interventions: Other: cancer cell lines establishment

INTERVENTIONS:
Other: cancer cell lines establishment — Detection of epithelial growth factor receptor (EGFR) mutation in malignant pleural effusion of lung cancer patients and cancer cell lines establishment
  Other Names: EGFR mutation; NSCLC cell line establishment

SUMMARY:
1. Detection EGFR mutation of cancer cells from malignant pleural effusion. 2. Established the cancer cell lines with without EGFR mutation from malignant pleural effusion.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of mortality in the world. Previous study has shown that about 88% lung cancer cases belong to non-small cell lung cancer (NSCLC) in Taiwan (1). Approximately 50~90% of NSCLC patients had expression (or described as overexpression) of EGFR in cancer (2,3). Although targeting the EGFR kinase domain using the inhibitors gefitinib (Iressa) and erlotinib (Tarceva) has no effect against solid tumors, it achieves impressive response in subgroup of NSCLC especially in Asian ethnic background, female sex, the absence of a history of smoking, and a tumor with histologic feature of adenocarcinoma (3,4,5). Molecular studies of highly responsive cases revealed high percentage of somatic mutation within the tyrosine kinase, ATP-binding domain of the EGFR gene (6). One possible explanation for this phenomenon is that the cancer cells are "addicted" to signaling via the mutant EGFRs and die when the mutant oncoprotein is inactivated (7). However, specific mechanisms underlying epidermal growth factor tyrosine kinase inhibitor (EGFR-TKI) induced cell death have not been well delineated (7).

Approximately 90% of mutations affect a few specific amino acids. In-frame deletions in exon 19 centered on codons 756 to 750 make up 45~50% of mutations, and another 35~45% consist of the missense mutation leucine to arginine at codon 858 (L858R) in exon 21 (8, 9, 10). The link between EGFR-TKI response and EGFR mutations have been confirmed, but the increased prevalence of mutations in Asian (25%to 50%) compared with North American and Western European patients (10%) is currently unexplained (6,8-12). The response rate to TKI treatment in mutations-positive is 77% (30% to 100% with most series >60%) compared with 10% in mutation-negative cases (6). It is interesting that exon 19 deletion have increased response and survival with TKIs compared with L858R cases (10, 13, 14). This is in contrast to the natural history of patients, where those with exon 19 deletions appear to have shorter survival than those with L858R (8). The biological difference is still unknown and different mutations may have different biochemical signaling properties (15).

In this study, we will collect the pleural effusion from lung cancer patients. We will characterize the EGFR status of the cancer cell from malignant pleural effusion and try to establish the cancer cell lines from these patients. We hope to establish several cell lines with different mutations and then we can compare the difference responses and signal pathways in these cell lines. We can also explore the detailed mechanism of TKI responsive cancer cell and try to develop other agent to enhance the pathways.

ELIGIBILITY:
Inclusion Criteria:

* All malignant pleural effusion related to NSCLC between April 2008 and March 2009.
* Older than 18 years old.
* The patients who received thoracentesis

Exclusion Criteria:

* The patients who are not compatible with inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
EGFR mutation in malignant pleural effusion of lung cancer patients cancer cell lines establishment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan